CLINICAL TRIAL: NCT04692233
Title: Qigong to Improve Frailty Among Older Cancer Survivors: A Randomized Controlled Trial
Brief Title: Qigong to Improve Frailty Among Older Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW19550
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Frailty; Survivorship; Elderly
Keywords: Qigong; Baduanjin; Cancer survivors; Frailty
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent statistician will generate the randomization list using computer and keep a secure copy of the randomization codes assignments. The group assignment will be sealed in separate opaque envelopes and centrally controlled. The BQ master and exercise trainer will not have knowledge about the aims of the study. The RAs responsible for assessing the outcomes and entering the data will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qigong (Experimental): The entire intervention will last 16 weeks, including 1-hour supervised training sessions twice a week during weeks 1 to 8 (training; 16 hours), and 1-hour supervised weekly follow-up sessions during weeks 9 to 16 (follow-up; 8 hours). The sessions will be supervised by an experienced qigong master. Throughout the intervention period, participants will be asked to self-practice BQ for 30 minutes twice a week from weeks 1 to 8, and then three times a week from weeks 9 to 16 (20 hours).
  Interventions: Behavioral: Qigong Baduanjin
- Light flexibility exercise (Active Comparator): The control group will practice light flexibility exercise without any abdominal breathing and meditation techniques. The duration and frequency of supervised sessions and self-practice will be identical to the qigong sessions. The supervised sessions will be conducted by a certified exercise trainer.
  Interventions: Behavioral: Light flexibility exercise

INTERVENTIONS:
Behavioral: Qigong Baduanjin — Qigong Baduanjin will comprise eight standardized movements. It is practiced as a combination of body movements, breath control, and mindful meditation, which is designed to improve qi function.
  Arms: Qigong
Behavioral: Light flexibility exercise — Each session will include seated and standing stretches that target upper (neck, arms, upper back, shoulders, back, and chest) and lower body (quadriceps, hamstrings, calves, and hips), as well as trunk rotations.
  Arms: Light flexibility exercise

SUMMARY:
The objective of the study is to examine the effects of a 16-week Baduanjin qigong intervention on frailty, physical performance, psychological well-being, and health-related quality of life (HRQoL) among post-treatment older cancer survivors. This will be a randomized controlled, assessor-blind trial conforming to the CONSORT guidelines. A total of 226 cancer survivors aged over 65 who have completed curative treatment and screened as pre-frail or frail will be recruited and randomized into intervention and control groups. It is expected that upon intervention completion, the intervention group will demonstrate greater reversed frailty status, more improvements in physical performance, better psychological well-being, and enhanced HRQoL compared to the control group. Study instruments will be Fried Phenotype Criteria, Edmonton Frail Scale, Short Physical Performance Battery, Geriatric Depression Scale, European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire, and a background questionnaire. The intervention comprises of 1-hour qigong group training twice a week for 8 weeks, then 1-hour weekly follow-up group practice for 8 weeks and self-practice. The control group participants will attend light flexibility exercise group sessions at the same duration and frequency as the intervention group. Intention-to-treat analysis will be performed.

DETAILED DESCRIPTION:
The number of cancer survivors is rising worldwide. For example, in the United States, the number of cancer survivors is projected to increase by 31%, from 16.9 million in 2019 to 22.2 million by 2030, of which two-thirds are aged 65 or above. Hong Kong is also facing a growing number of cancer survivors, especially in older adults, due to advances in early detection and treatments and an aging population. The Hong Kong Cancer Strategy 2019 launched by the Hong Kong Government and Hospital Authority seeks to enhance cancer survivorship and surveillance management.

Older cancer survivors, making up the majority of survivors, tend to suffer from the combined effect of aging and long-term impacts of cancer, resulting in higher morbidity rates and poorer health-related quality of life than older adults without a cancer history. Tailored care for survivorship in older adults with cancer is highly important to reduce healthcare and economic burdens. In geriatric oncology, frailty status is an emerging health indicator with prognostic value. Nearly 80% of older cancer survivors have pre-frailty and frailty status that is linked to adverse health outcomes such as disability, impaired quality of life, falls, and death. There is a tremendous need to develop effective lifestyle interventions to reverse frailty status in the older cancer survivors. However, many clinical trials exclude participants older than 65 years old, and in real-world practice, many clinicians and policymakers advocate lifestyle modifications for older survivors less frequently than for younger survivors. The proposed project responds to an urgent research agenda in cancer survivorship that calls for interventions for addressing frailty.

The primary aim of this study is to evaluate the effect of a 16-week Baduanjin intervention on reversing frailty status among pre-frail and frail older cancer survivors. Reversal of frailty status is expected to be accompanied by improvements in patients' functioning, psychological well-being, and quality of life, and can reduce health service utilization and healthcare costs. Baduanjin is a simple form of qigong and can be performed by participants as and when needed after appropriate training. If the intervention proves effective, the widespread incorporation of qigong into treatment recommendations for cancer survivors can be easily translated into practice with little healthcare professional or patient burden.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥65
2. diagnosed with stage I-III non-metastatic cancer
3. completed primary treatment with curative intent (surgery, chemotherapy, and/or radiation therapy) 6 months to 5 years prior to baseline assessments with no recurrence or occurrence of additional cancers
4. classified as pre-frail or frail based on Fried frailty criteria
5. can communicate in Cantonese or Putonghua
6. written informed consent

Exclusion Criteria:

1. regular qigong training or other mind body intervention (once or more per week) within the previous 6 months
2. medical conditions affecting mobility, predisposing to falls, or precluding qigong practice (e.g., neurological disease, musculoskeletal disorder, recent myocardial infarction, breathing difficulties requiring oxygen)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 226 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Improvement in frailty status | at study entry, post-training, post-intervention, 6 months post intervention, 12 months post intervention
  Participants' frailty status will be assessed using the Fried frailty criteria, which consists of 5 criteria: slowness , weakness , unintentional weight loss , exhaustion and low activity. Patients with no criteria are considered robust, patients with 1 or 2 criteria are considered pre-frail, and patients with ≥3 criteria are considered frail.

SECONDARY OUTCOMES:
Improvement in frailty scores | at study entry, post-training, post-intervention, 6 months post intervention, 12 months post intervention
  The Edmonton Frail Scale will be used to capture changes in frailty as a continuous score. As a multidimensional view, it will complement the physical-based Fried criteria regarding the intervention effect. The scale consists of 11 items, which cover nine domains (cognition, general health status, functional independence, social support, medication use, nutrition, mood, continence, and functional performance). The higher total scores represent more severe frailty states.
Physical performance | at study entry, post-training, post-intervention, 6 months post intervention, 12 months post intervention
  Short Physical Performance Battery is an objective assessment tool used to measure the physical performance of participants in three functional tasks.
Psychological well-being | at study entry, post-training, post-intervention, 6 months post intervention, 12 months post intervention
  The Short-Form Geriatric Depression Scale (15 items) will be used to measure psychological well-being. Scores range from 0 to 15, with higher scores representing more severe depressive symptoms.
Health-related quality of life | at study entry, post-training, post-intervention, 6 months post intervention, 12 months post intervention
  European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire-C30 (30 items) will be used to assess health-related quality of life specifically in cancer patients. The questionnaire is composed of five functional scales, three symptom scales, a global health status / QoL scale, and six single items. scale. Scores of all subscales and single-item measures range from 0 to 100. Higher scores for functional scales represent higher level of functioning, global health status/quality of life, but higher scores for a symptom scale / item represent a higher level of symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Shuk Ting Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request as decided by the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 3 years after the manuscript on main findings is published.